CLINICAL TRIAL: NCT06347640
Title: The Outcome of Pulp Revascularization of Necrotic Mature Permanent Teeth With Periapical Lesion Using Platelet-rich Fibrin Versus Induced Bleeding: Randomized Clinical Trial
Brief Title: Outcome of Pulp Revascularization of Necrotic Mature Permanent Teeth Using Platelet-rich Fibrin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lama Awawdeh, Professor, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KingAbdullahUH2
Record Dates: First submitted 2024-03-23; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Pulp Revascularization

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induced bleeding group (Active Comparator): revascularization of mature necrotic permanent teeth treated by induced bleeding though apex of the tooth
  Interventions: Biological: induced bleeding
- Platelet-rich fibrin (PRF) group (Experimental): revascularization of mature necrotic permanent teeth treated using platelet-rich fibrin (PRF)
  Interventions: Biological: plasma rich fibrin

INTERVENTIONS:
Biological: induced bleeding — revascularization of tooth is achieved by induced bleeding
  Arms: Induced bleeding group
Biological: plasma rich fibrin — revascularization of tooth is achieved by plasma rich fibrin
  Arms: Platelet-rich fibrin (PRF) group

SUMMARY:
Regenerative endodontic procedures are intended to replace damaged tooth structures, including dentine and root structures, in addition to cells of the pulp-dentine complex. This treatment modality have been tested on immature necrotic teeth because they are anticipated to have a greater chance of pulp tissue regeneration.

However, it has been recently suggested for treating fully formed mature necrotic permanent teeth with closed apices since the conventional root canal treatment yielded many drawbacks.

A number of studies have evaluated the regeneration outcomes of using blood clot as a scaffold. However, there are limited studies in the literature on using other scaffolds such as platelet-rich fibrin (PRF).

This clinical study will evaluate clinically and radiographically the effectiveness of PRF versus induced bleeding in treating mature necrotic teeth. Fifty patients with necrotic mature teeth with periapical lesions will be invited to participate in this study. Teeth will be treated using calcium hydroxide as intracanal medicament then using PRF (n=25) and blood clot (n=25) as scaffold. All teeth will be sealed coronally using NeoMTA Plus™. Treated teeth will be assessed clinically and radiographically using 2D periapical radiographs. The reported clinical and radiographic outcomes will be compared using SPSS.

DETAILED DESCRIPTION:
The regeneration procedures have been focused on immature teeth since there is a need for a treatment modality to give a chance for root maturation, apical closure, and root canal walls thickening which cannot be achieved by other procedures like apexification. Immature teeth have a greater chance of pulp tissue regeneration. The presence of an open apex will allow the stem cells from the apical papilla to migrate into root canals.

In the case of mature teeth, the presence of complex anatomy causes difficulties in disinfection. In addition, the presence of narrow apical pathway for stem cells migration makes them weak candidates for regeneration. However, the use of conventional root canal therapy has many drawbacks.

A retrospective study reported that even though conventional root canal therapy had prolonged tooth survival, pulp removal still led to tooth loss in comparison with teeth with normal pulp. Losing the pulp means reduced levels of proprioception in addition to the innate immunity that is disallowed after root canal therapy leaving remaining bacterial colonies in the root canal system. By applying regeneration techniques in mature teeth, we have the chance to avoid the previously mentioned drawbacks of root canal therapy and restore the neurovascular system with immune cells that will act as a line of defense mechanism against microbial attacks.

A few studies and case reports have investigated the effectiveness of regeneration procedures using blood clot as a scaffold in treating mature necrotic teeth. The idea that led toward the use of platelet concentrates as a scaffold was that concentrated platelets and growth factors collected in plasma solutions could promote local healing. Comparing it to blood clot, it increased cell proliferation over time due to its increased concentration of growth factors.

Given the drawbacks of conventional root canal treatment and limited studies in the literature on using other treatment modalities in treating mature necrotic teeth, hence the need for a randomized clinical trial with large sample size and long follow-ups emerge. This clinical study will evaluate clinically and radiographically the effectiveness of PRF versus induced bleeding in treating mature necrotic teeth.

ELIGIBILITY:
Inclusion Criteria

1. Anterior or posterior mature tooth diagnosed with necrotic pulp in the presence of a periapical lesion,
2. Pulp space is not needed for post and core restoration.
3. Patients are not allergic to the medicaments necessary to complete the procedure.

Exclusion Criteria

1. Medically compromised patient.
2. Patient with generalized chronic periodontitis.
3. Teeth with previous root canal treatment.
4. Periodontal pocket larger than 3mm.
5. Teeth with vertical fractures
6. Non-restorable teeth

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete healing | treated teeth will be evaluated from start of intervention up to 100 months
  Assess clinically and radiographically absence of symptoms and signs And evidence for continuation of root development after regeneration procedures

SECONDARY OUTCOMES:
regain the pulp sensibility | pulp sensibility will be evaluated one year after treatment
  asses pulp sensibility using cold test

CONTACTS AND LOCATIONS:
Overall Officials: Lama Awawdeh, Study Chair — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No